CLINICAL TRIAL: NCT00352313
Title: A Phase I/II Study of ATN-161 and Carboplatin in Adult Patients With Recurrent Intracranial Malignant Glioma
Brief Title: ATN-161 and Carboplatin in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 060170; 06-C-0170; NCI-P6790; ATN-161-002; CDR0000487605; NCT00340041 (obsolete NCT alias)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult gliosarcoma; adult mixed glioma; adult anaplastic astrocytoma; recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Gliosarcoma; Glioma; Astrocytoma; Brain Neoplasms; Glioblastoma | interventions — acetyl-prolyl-histidyl-seryl-cysteinyl-asparaginamide; Carboplatin

ARMS (2):
- Phase I (Experimental): Patients receive ATN-161 IV over 10 minutes 3 times weekly in weeks 1-6 and carboplatin IV over 20 minutes in week 3 during course 1. Beginning in course 2, patients receive carboplatin IV over 20 minutes in week 1 and ATN-161 IV over 10 minutes 3 times weekly in weeks 1-4. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ATN-161; Drug: carboplatin
- Phase II (Experimental): Patients receive carboplatin IV in week 1 and ATN-161 IV, at the MTD determined in phase I, 3 times weekly in weeks 1-4. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ATN-161; Drug: carboplatin

INTERVENTIONS:
Drug: ATN-161 — Given IV
Drug: carboplatin — Given IV

SUMMARY:
RATIONALE: ATN-161 may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving ATN-161 together with carboplatin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ATN-161 when given together with carboplatin and to see how well they work in treating patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the safety of ATN-161 and carboplatin in patients with recurrent intracranial malignant glioma.
* Determine the maximum tolerated dose of ATN-161 when administered with carboplatin in these patients. (phase I)
* Determine the antitumor activity of ATN-161 when administered with carboplatin in these patients. (phase II)

Secondary

* Describe the effects of this regimen on potential biomarkers of activity, including functional imaging with brain perfusion scans and circulating endothelial progenitor cells.
* Obtain preliminary evidence of efficacy of this regimen in these patients. (phase I)
* Characterize the plasma concentrations of this regimen in these patients. (phase I)

OUTLINE: This is an open-label, phase I dose-escalation study of ATN-161 followed by a phase II study. Patients in the phase II portion of the study are stratified according to tumor type (glioblastoma multiforme vs anaplastic glioma).

* Phase I: Patients receive ATN-161 IV over 10 minutes 3 times weekly in weeks 1-6 and carboplatin IV over 20 minutes in week 3 during course 1. Beginning in course 2, patients receive carboplatin IV over 20 minutes in week 1 and ATN-161 IV over 10 minutes 3 times weekly in weeks 1-4. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ATN-161 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity during the first 6 weeks of treatment.

* Phase II: Patients receive carboplatin IV in week 1 and ATN-161 IV, at the MTD determined in phase I, 3 times weekly in weeks 1-4. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and then periodically during phase I course 1 for pharmacokinetic and pharmacodynamic analysis and at baseline and then periodically during study for biomarker (e.g., circulating endothelial progenitor cells) correlative studies.

After completion of study treatment, patients are followed for 28 days.

PROJECTED ACCRUAL: A total of 82 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial malignant glioma

  * Original low-grade glioma histology allowed provided there is subsequent histologic confirmation of malignant glioma
* Any of the following diagnoses:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
* Recurrent disease

  * Must have failed prior radiotherapy

    * Must have confirmation of true progressive disease (rather than radiation necrosis) based upon either positron emission tomography or thallium scanning, MR spectroscopy, or surgical documentation of disease if radiographic recurrence is within the high-dose radiation field (for patients who underwent prior interstitial brachytherapy or stereotactic radiosurgery)
* Prior recent resection of recurrent or progressive tumors allowed if all of the following criteria are met:

  * Recovered from prior surgery
  * Evaluable disease after resection
* Unequivocal evidence of tumor progression by MRI

  * Steroid dose must be stable for ≥ 5 days prior to MRI

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 8 weeks
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* AST < 2.5 times upper limit of normal (ULN)
* Bilirubin < 2.5 times ULN
* Creatinine < 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study treatment
* No significant medical illness that would preclude study treatment
* No history of other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix) unless disease is in complete remission and off all therapy for ≥ 1 year
* No active infection or serious intercurrent medical illness
* No disease that will obscure toxicity or dangerously alter drug metabolism
* Able to undergo MRI scan and receive contrast agents for perfusion scanning

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 28 days since prior cytotoxic therapy
* At least 14 days since prior vincristine
* At least 42 days since prior nitrosoureas
* At least 21 days since prior procarbazine
* At least 7 days since prior interferon, tamoxifen, thalidomide, isotretinoin, or other noncytotoxic agents (radiosensitizer does not count)
* At least 14 days since prior noncytotoxic investigational agents
* At least 42 days since prior radiotherapy
* No prior cisplatin, carboplatin, oxaliplatin, or platinum-containing analogue
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* No other concurrent anticancer therapy (including chemotherapy, radiotherapy, hormonal therapy, or immunotherapy)
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety
Maximum tolerated dose (phase I)
Progression-free survival at 6 months
Response rate (phase I)
Overall survival

SECONDARY OUTCOMES:
Efficacy
Response rate (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Fine, MD, Principal Investigator — NCI - Neuro-Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States